CLINICAL TRIAL: NCT05751161
Title: Effect of Gait Training With Auditory Stimuli on Dynamic Balance, Gait and Functional Independence in Chronic Stroke
Brief Title: Effect of Gait Training With Auditory Stimuli on Balance, Gait & Funtional Independence in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0211
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- effect of gait training with AS on dynamic balance, gait and functional independence in stroke (Experimental): Patients with chronic stroke receive gait training with auditory stimuli to improve dynamic balance, gait and functional independence.
  Interventions: Other: conventional gait training
- effect of conventional gait training on dynamic balance, gait and functional independence in stroke (Other): Patients in this group receive conventional gait training only to improve dynamic balance, gait and functional independence .Patients did not receive auditory stimuli for gait training.
  Interventions: Other: conventional gait training

INTERVENTIONS:
Other: conventional gait training — The experimental group received circuit gait training with auditory stimuli using a smartphone metronome application. The training program consisted of eight different activities i.e. tandem walk, one-leg standing, military march, sitting up and forward walk, lateral walk, kicking a ball towards the wall, walking on a set pattern and obstacle walk .Patient will practice each task for 3-4 mints and three times per week.
  Other Names: Gait training with auditory stimuli

SUMMARY:
To determine the effect of gait training with auditory stimuli on dynamic balance, gait and functional independence on chronic stroke.

DETAILED DESCRIPTION:
The purpose of this study is to find the effect of gait training with auditory stimuli using a smart phone metronome application on dynamic balance, gait and functional abilities of chronic stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* both gender
* Age between 30-70
* More than 6 months after the stroke
* Able to walk more than 10 meters independently
* MMSE score of 24

Exclusion Criteria:

* Dependent gait
* Aphasia
* Any hearing or visual defects
* Moderate to severe cognitive disorder
* People not willing to participtae

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 6 weeks
  To identify the effect of treatment on dynamic balance. The BBS consists of 14 items scored on a 5 point ordinal scale , ramging from 0-4 ..0 means unable to sit without support .4 means able to sit independently.

SECONDARY OUTCOMES:
Barthel index | 6 weeks
  it is an ordinal scale that measures functional independence in the domain of personal care and mobility.
Gait speed | 6 weeks
  it is the time one takes to walk a specific distance on level surface over a short distance. A distance of 3 to 10 meters is measured over a level surface with 2 meters acceleration and 2 meter for decleration
POMA | 6 weeks
  It evaluates dynamic balance and walking patters.

CONTACTS AND LOCATIONS:
Overall Officials: maria samad, Principal Investigator — Riphah International University; fatima tariq, Principal Investigator — Riphah International University
Locations (1):
- Pakistan society for the rehabilitation of disabled, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Park MH, Won JI. The effects of task-oriented training with altered sensory input on balance in patients with chronic stroke. J Phys Ther Sci. 2017 Jul;29(7):1208-1211. doi: 10.1589/jpts.29.1208. Epub 2017 Jul 15. PMID 28744049